CLINICAL TRIAL: NCT01506375
Title: Safety, Clinical Tolerability and Immunogenicity of gpASIT+TM Administered Subcutaneously to Hay Fever Patients Either Alone or in Presence of DnaK Immunoregulating Adjuvant
Brief Title: Safety of gpASIT+TM Subcutaneously Administered to Hay Fever Patients With or Without Immunoregulating Adjuvant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioTech Tools S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: gpASIT006; 2011-004486-33 (EudraCT Number)
Record Dates: First submitted 2011-12-07; First posted 2012-01-10 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2012-08

CONDITIONS: Hay Fever
Keywords: seasonal allergic rhinoconjunctivitis; grass pollen; allergen specific immunotherapy
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- gpASIT (Experimental): grass pollen peptides alone
  Interventions: Biological: gpASIT+TM
- gpASIT/adjuvant (Experimental): grass pollen peptides + adjuvant
  Interventions: Biological: gpASIT+TM + adjuvant

INTERVENTIONS:
Biological: gpASIT+TM — 1 subcutaneous injection every 7 days during 29 days
  Arms: gpASIT
Biological: gpASIT+TM + adjuvant — 1 subcutaneous injection every 7 days during 29 days
  Arms: gpASIT/adjuvant

SUMMARY:
The aim of the study is to compare the safety, clinical tolerability, immunogenicity and efficacy of gpASIT+TM (grass pollen peptides) alone and combined with an immunoregulating adjuvant, in a short course administration (5 injections over 4 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Subject has given written informed consent
* Age between 18 and 50 years
* The subjects are in good physical and mental health according to his/her medical history, vital signs, and clinical status
* Male or non-pregnant, non-lactating female
* Females unable to bear children must have documentation of such in the CRF (i.e. tubule ligation, hysterectomy, or post-menopausal (defined as a minimum of one year since the last menstrual period))
* Allergy diagnosis:

  * A medical history of moderate to severe seasonal allergic rhinoconjunctivitis (SAR) during the grass pollen season during at least the two previous years
  * A positive skin prick test (wheal diameter ≥ 3 mm) to grass-pollen mixture
  * Specific IgE against grass pollen (IgE > 0.7 kU/l) [using recombinant mixture of rPhl p1 and rPhl p5b Phleum pratense (g213)]
* Subjects never treated by immunotherapy or subjects for whom the immunotherapy ended at December 31, 2009 and who had as well moderate to severe symptoms in the two previous years (2010 and 2011)

Exclusion Criteria:

* Subjects with current immunotherapy and subjects who underwent a previous immunotherapy within the last 2 years
* Participation in another clinical trial and/or treatment with an experimental drug within the last 3 months
* A history of hypersensitivity to the excipients of investigational products
* Subjects with perennial asthma (regular intake of inhaled corticosteroids outside the pollen season: consumption on a daily base or patients who are taking a reliever more than twice a week)
* Subjects with severe seasonal asthma requiring long acting beta agonist AND inhaled steroid treatment
* Subjects with a VC < 80% and a FEV1 < 70% of predicted value at the screening visit
* Subjects symptomatic to perennial inhalant allergens who should need antihistamine drug or systemic corticoids to relieve allergic symptoms during the treatment period
* Subjects with documented evidence of chronic sinusitis (as determined by Investigator)
* Subjects with rhinitis medicamentosa, non-specific rhinitis (to food dye, preservative agent…)
* Subjects with a history of renal disease or chronic hepatic disease
* Subject with malignant disease, autoimmune disease
* Any chronic disease, which may impair the subject's ability to participate in the trial
* Subjects requiring beta-blockers medication
* Chronic use of concomitant medications that would affect assessment of the effectiveness of the trial medication (e.g. tricyclic antidepressants)
* Regular consumption of corticoids (oral, topic or nasal) or of anti-histaminic drugs within 4 weeks preceding the trial (screening visit)
* Any consumption of corticoids (oral, topic or nasal) or of anti-histaminic drugs within 1 week preceding the trial (screening visit)
* Subject with febrile illness (> 37.5°C, oral)
* A known positive serology for HIV-1/2, HBV or HCV
* Subjects that are immunocompromised by medication or illness, have received a vaccine, corticoids or immunosuppressive medications within 1 month before trial entry
* Receipt of blood or a blood derivative in the past 6 months preceding trial entry
* Female subjects who are pregnant, lactating, or of child-bearing potential and not protected from pregnancy by a sufficiently reliable method
* Any condition which could be incompatible with protocol understanding and compliance
* Subjects who have forfeited their freedom by administrative or legal award or who are under guardianship
* Unreliable subjects including non-compliant subjects, subjects with known alcoholism or drug abuse or with a history of a serious psychiatric disorder as well as subjects unwilling to give informed consent or to abide by the requirements of the protocol
* Subjects without means of contacting the Investigator rapidly in case of emergency, or not able to be contacted rapidly by the Investigator

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-11; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Safety of the treatment | up to the end of the grass pollen season
  Safety will be evaluated by the following parameters: general physical status, vital signs, haematological parameters, general biochemical parameters, solicited local adverse events, all (serious) adverse events, immunological analysis (total IgG and IgE), inflammatory parameters (CRP) and anti-adjuvant mmunoglobulins.
Clinical tolerability of the treatment | Duration of treatment period (4 weeks)
  The clinical tolerability will by assessed through the solicited local adverse events, all (serious) adverse events and the investigator and subject opinion.

SECONDARY OUTCOMES:
Impact of gpASIT+TM with or without adjuvant on the immunological status of the subjects. | up to 1 year after the start of treatment
  The following parameters will be assessed: allergen-specific immunoglobulins and blocking antibodies.
Impact of gpASIT+TM with or without adjuvant on the grass pollen allergic symptoms of the subjects. | During the pollen season
  The following parameters will be recorded: symptom and rescue medication scores (diary cards), Quality-of-Life (RQLQ(S)).
Long-term follow-up of the patients | 1 year after the start of treatment
  Safety parameters will be: immunological analysis (Total IgG and IgE), inflammatory parameters (CRP), DnaK-specific immunoglobulins and SAEs.
  Immunogenicity parameters will be: evolution of grass pollen specific immunoglobulins and of blocking antibodies.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitaire Ziekenhuis van Leuven, Leuven, Belgium